CLINICAL TRIAL: NCT07172789
Title: Head dOwn Position Before Endovascular Treatment for Large veSsel Occlusion (HOPES5): a Prospective, Randomized, Open Label, Blinded-end Point, Multi-center Study
Brief Title: Head dOwn Position Before Endovascular Treatment for Large veSsel Occlusion (HOPES5)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Director, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Y (2025) 320
Record Dates: First submitted 2025-09-02; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Head-Down Tilt

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HDP (Experimental): the HDP group receive -20° Trendelenburg prior endovascular treatment.
  Interventions: Other: head down position
- Control (No Intervention)

INTERVENTIONS:
Other: head down position — the patient is positioned at a -20° Trendelenburg
  Other Names: Trendelenburg
  Arms: HDP

SUMMARY:
Recent studies suggest that head-down positioning (HDP) intervention may improve outcomes in ischemic stroke. In the era of reperfusion therapy, a key protective strategy is to administer neuroprotective interventions before recanalization to reduce the loss of the ischemic penumbra, thereby salvaging more penumbral tissue after revascularization and ultimately improving clinical outcomes. Based on this concept, and considering the neuroprotective effects of HDP, the investigators hypothesize that HDP intervention prior to endovascular therapy (EVT) in patients with large vessel occlusion could improve clinical outcomes. This hypothesis is further supported by a recent clinical study (NCT03728738), which demonstrated that compared to a sitting up position (30°), a flat supine position (0°) before EVT significantly reduced the incidence of neurological deterioration prior to the procedure. Building on the above rationale, this trial aims to investigate the efficacy and safety of HDP intervention prior to EVT in patients with large vessel occlusion.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Patients with acute large vessel occlusion scheduled for endovascular thrombectomy within 24 hours of symptom onset;
* Baseline National Institute of Health Stroke Scale (NIHSS) ≥ 6;
* Expected waiting time from randomization to femoral artery puncture is more than 30 minutes;
* ASPECTS/pc-ASPECTS score ≥ 6 on baseline non-contrast CT or DWI;
* Modified Rankin Scale score before stroke onset ≤ 1;
* Signed informed consent by patient or their legally authorized representative.

Exclusion Criteria:

* Hemorrhagic stroke: cerebral hemorrhage, subarachnoid hemorrhage;
* Severe hepatic or renal dysfunction, increase in ALT or AST (more than 2 times of upper limit of normal value), increase in serum creatinine (more than 1.5 times of upper limit of normal value) or requiring dialysis;
* Severe hypertension before randomization (systolic blood pressure >185 mmHg or diastolic blood pressure >110 mmHg);
* Cardiac insufficiency (NYHA Class ≥II);
* Pregnancy, plan to get pregnant or during lactation;
* Patients at significant risk of aspiration (e.g., obvious nausea and vomiting);
* The estimated life expectancy is less than 6 months due to other serious diseases;
* Other conditions unsuitable for this clinical study assessed by researcher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
early neurologic improvement (ENI) | 24±8 hours
  ENI was defined as more than 4-point decrease in NIHSS within 24±8 hours;

SECONDARY OUTCOMES:
proportion of good collateral circulation status | during the first angiography examination
  good collateral circulation status was defined as ASITN/SIR grade 3-4.
Change in National Institutes of Health Stroke Scale (NIHSS) | Immediately before endovascular treatment
  the minimum and maximum values of NIHSS are 0 and 42, respectively; higher NIHSS mean a worse outcome.
Change in National Institutes of Health Stroke Scale (NIHSS) | 24±8 hours
  the minimum and maximum values of NIHSS are 0 and 42, respectively; higher NIHSS mean a worse outcome.
Changes in cerebral infarct volume | 24±8 hours
  infarct volume was measured by MRI-DWI
Changes in cerebral edema | 24±8 hours
  change in cerebral edema was measured based on middle shift on CT or MRI
Change in National Institutes of Health Stroke Scale (NIHSS) | 10±2 days
  the minimum and maximum values of NIHSS are 0 and 42, respectively; higher NIHSS mean a worse outcome.
proportion of modified Rankin Scale (mRS) 0-1 | 90±7 days
  The minimum and maximum values of mRS are 0 and 6, respectively; higher score mean a worse outcome
proportion of modified Rankin Scale (mRS) 0-2 | 90±7 days
  The minimum and maximum values of mRS are 0 and 6, respectively; higher score mean a worse outcome
ordinal distribution of modified Rankin Scale (mRS) | 90±7 days
  The minimum and maximum values of mRS are 0 and 6, respectively; higher score mean a worse outcome
new stroke or other vascular event(s) | 90±7 days
percentage of severe adverse events | 24±8 hours
proportion of symptomatic intracranial hemorrhage | 24±8 hours
  symptomatic intracranial hemorrhage is defined as a NIHSS increase ≥4 caused by intracranial hemorrhage
proportion of intraparenchymal hemorrhage (PH) | 24±8 hours
  PH was defined as confluent bleeding occupying and causing mass effect
all-cause mortality | 10±2 days

OTHER OUTCOMES:
changes in dynamic cerebral autoregulation (dCA) | 24±8 hours
  dCA data include phase difference (the main parameter, determined as the phase shift angle ranging from 0° to 90°), gain (difference in the amplitude between CBFV and ABP), and the coherence function (indicates signal-to-noise ratio), which is determined according to previous report (Guo ZN, Guo WT, Liu J, et al. Changes in cerebral autoregulation and blood biomarkers after remote ischemic preconditioning.)
changes in cortical oxygen saturation | 24±8 hours
  cortical oxygen saturation is determined by near infrared spectroscopy
changes in serum biomarkers | 24±8 hours
  serum biomarkers include MMP-9, TNF-alpha, IL-1beta, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Hui-Sheng Chen, Shenyang, None Selected, China

IPD SHARING:
Plan to Share IPD: Undecided